CLINICAL TRIAL: NCT03625531
Title: A Multicenter Randomized Trial of Personalized Acupuncture, Fixed Acupuncture, Letrozole and Placebo on Live Birth for Infertility in Women With Polycystic Ovary Syndrome
Brief Title: A Trial of Personalized Acupuncture, Fixed Acupuncture, Letrozole and Placebo on Live Birth in Women With PCOS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hongxia Ma (Other)
Responsible Party: Sponsor-Investigator, Hongxia Ma, professor, The First Affiliated Hospital of Guangzhou Medical University
Organization: The First Affiliated Hospital of Guangzhou Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PPCOSAct
Record Dates: First submitted 2018-07-13; First posted 2018-08-10 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Acupuncture; Polycystic Ovary Syndrome; Personalized protocol; Fixed protocol; Letrozole
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Acupuncture Therapy; Letrozole

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Personalized acupuncture (Experimental): Two sets of acupoints will be selected for the two types. The basic acupoint-prescription includes CV 4, CV 6, CV 12 and SP 6 bilaterally, ST 25 bilaterally, EX-CA 1 bilaterally, ST 40 bilaterally and SP 9 bilaterally. Additional point ST 36 bilaterally and moxibustion as adjuvant therapy will be added for the type of yang deficiency of spleen and kidney, while additional points K 13, LR 3 for the type of yin deficiency of liver and kidney. Besides, flexible modifications of 2-3 acupoints will be performed according to patients special symptoms.
  Interventions: Other: Acupuncture
- Fixed acupuncture (Experimental): Two sets of acupuncture points will be alternated every second treatment. The first set consists of CV 3, CV 6, ST 29 bilaterally, SP 6 bilaterally, SP 9 bilaterally, GV 20 and LI 4 bilaterally. The second set consists of 13 needles: ST 25 bilaterally, ST 29 bilaterally, CV 3, CV 6, SP 6 bilaterally, LR 3 bilaterally, PC 6 bilaterally and GV 20. The following points will be connected to an electrical stimulator: ST 25 bilaterally, ST 29 bilaterally, SP 6 bilaterally, LR 3 bilaterally.
  Interventions: Other: Acupuncture
- Letrozole (Active Comparator): Women in the letrozole group will be given letrozole (Femara, Novartis Pharmaceuticals, Basel, Switzerland) from day 3 to day 7 of the spontaneous menstrual cycle or after a withdrawal bleeding following progestin. The maximum daily dose of letrozole will be 7.5 mg (3 pills) daily for five days.
  Interventions: Drug: Letrozole
- Placebo letrozole (Placebo Comparator): Women will receive placebo letrozole with no acupuncture from day 3 to day 7 of the spontaneous menstrual cycle or after a withdrawal bleeding following progestin. Placebo letrozole will be given in the same way as letrozole.
  Interventions: Drug: Placebo letrozole

INTERVENTIONS:
Other: Acupuncture — Women in both personalized and fixed acupuncture groups will receive acupuncture treatment three times a week. Acupuncture treatment will start on day 3 after a spontaneous period or after a withdrawal bleeding following progestin. Each treatment session will last for 30-60 minutes, with a maximum of 48 treatment sessions over 16 weeks. If they become pregnant, the acupuncture treatment will be stopped. For personalized and fixed acupuncture group, credibility and expectancy questionnaires will be completed on the third acupuncture treatment and the last acupuncture treatment.
  Arms: Fixed acupuncture; Personalized acupuncture
Drug: Letrozole — Letrozole will be started on day 3 to day 7 of the spontaneous period or a withdrawal bleeding following progestin. If there is response with ovulation, this dose will be maintained. In those with no ovulatory response, letrozole tablets of the next ovulation cycle will be take on the day 28 of the menstrual cycle and the letrozole dose will be increased to 5 mg (2 pills) a day for 5 days. If there is still no response, the dose will be increased to 7.5 mg per day for 5 days in the next cycle. The maximum daily dose of letrozole will be 7.5 mg (3 pills) daily for five days.
  Other Names: Femara, Novartis Pharmaceuticals
  Arms: Letrozole
Drug: Placebo letrozole — Placebo letrozole will be given in the same way as letrozole. Women will receive 1 tablet a day of placebo letrozole from the day 3 to day 7 of the menstrual cycle and placebo letrozole dose will be increased 2 tablets a day in the next cycle if there is no response. The maximum daily dose of placebo letrozole will be 3 tablets daily for five days.
  Other Names: Placebo
  Arms: Placebo letrozole

SUMMARY:
This study is a randomized assessor-blind controlled trial. A total of 1,100 women with PCOS will be recruited from 28 hospitals and randomly allocated into four groups: personalized acupuncture, fixed acupuncture, letrozole or placebo letrozole. Patients will receive treatment for 16 weeks and the primary outcome is live birth.

DETAILED DESCRIPTION:
Traditional Chinese Medicine (TCM) usually involves syndrome and disease differentiation, and for acupuncture selection of appropriate points and skillful needling techniques. Many clinical trials on acupuncture used fixed acupuncture protocols without accounting for individual differences. We here design a multicenter randomized controlled trial to evaluate whether personalized or fixed acupuncture increases the likelihood of live births for infertility in women with polycystic ovary syndrome (PCOS) compared with letrozole or placebo letrozole. We hypothesis that letrozole is more effective than personalized acupuncture and that personalized acupuncture is more effective than standardized acupuncture, which is more effective than placebo letrozole.

ELIGIBILITY:
Inclusion criteria

1. Age of women between 20 and 40 years.
2. Chronic oligomenorrhea or amenorrhea: oligomenorrhea is defined as an intermenstrual interval > 35 days or < 8 menstrual bleedings in the past year. Amenorrhea is defined as an intermenstrual interval >90 days.
3. Hyperandrogenism (either hirsutism or hyperandrogenemia) or polycystic ovaries on ultrasound. Hirsutism is determined by a modified Ferriman-Gallwey Score ≥ 5 at screening examination, and biochemical hyperandrogenism is defined as total testosterone (T) > 2.6 nmol/L and free testosterone ≥ 6.0 pg/mL. Polycystic ovaries are present when there are ≥ 12 antral follicles (2 - 9 mm) or ovarian volume > 10 mL on transvaginal scanning.
4. At least one patent tube shown by hysterosalpingogram or diagnostic laparoscopy within 3 years if the patient does not have a history of abortion or pelvic operation. If the patient has a history of pregnancy and no history of pelvic operation within the past 5 years, she is not required to undergo a tubal patency test.
5. Sperm concentration ⩾ 15 × 106/mL and total motility ⩾ 40% or total motile sperm count ⩾ 9 million in the semen analysis of the husband. Agree to have regular intercourse i.e. 2-3 times per week during the study period.

Exclusion criteria

1. Exclusion of other endocrine disorders: a. patients with hyperprolactinemia (defined as two prolactin levels at least one week apart ≥ 25 ng/mL); b. Patients with FSH levels > 15 mIU/mL. A normal level within the last year is adequate for entry; c. Patients with uncorrected thyroid disease (defined as TSH < 0.2 mIU/mL or > 5.5 mIU/mL). A normal level within the last year is adequate for entry. d. Patients diagnosed with Type I or Type II diabetes who are poorly controlled (defined as HbA1c level > 7.0%), or patients receiving antidiabetic medications such as metformin, insulin, thiazolidinediones, acarbose, or sulfonylureas. e. Patients with suspected Cushing's syndrome.
2. Use of other TCM treatments including Chinese herbal prescriptions and acupuncture in the past 3 months.
3. Use of other western medications known to affect reproductive function or metabolism in the past 2 months.
4. Pregnancy within the past 6 weeks.
5. Within 6 weeks postabortion or postpartum.
6. Breastfeeding within the last 6 months.
7. Not willing to give written consent to the study.
8. Additional exclusion criteria are as follows.

   1. Patients taking other medications known to affect reproductive function or metabolism. These medications include oral contraceptives, depot progestins, hormonal implants (including Implanon), GnRH agonists and antagonists, antiandrogens, gonadotropins, antiobesity drugs, antidiabetic drugs such as metformin and thiazolidinediones, somatostatin, diazoxide, angiotensin-converting-enzyme (ACE) inhibitors, and calcium channel blockers. The washout period on these medicationswill be two months, longer washouts may be necessary for certain depot contraceptive forms or implants, especially where the implants are still in place. A one-month washout will be required for patients on depot progestins.
   2. Patients with liver disease defined as AST or ALT > 2 times normal or total bilirubin > 2.5 mg/dL. Patients with renal disease defined as BUN > 30 mg/dL or serum creatinine > 1.4 mg/dL.
   3. Patients with hemoglobin < 10 g/dL.
   4. Patients with a history of deep venous thrombosis, pulmonary embolus, or cerebrovascular accident.
   5. Patients with known heart disease that is likely to be exacerbated by pregnancy.
   6. Patients with a history of, or suspected cervical carcinoma, endometrial carcinoma, or breast carcinoma. A normal Pap smear result will be required for women 21 and over.
   7. Patients with a current history of alcohol abuse. Alcohol abuse is defined as >14 drinks/week or binge drinking.
   8. Patients enrolled into other investigative studies that require medications, prescribe the study medications, limit intercourse, or otherwise prevent compliance with the protocol.
   9. Patients who anticipate taking longer than a one-month break during the protocol should not be enrolled.
   10. Patients with a suspected adrenal or ovarian tumor secreting androgens.
   11. Couples with previous sterilization procedures (vasectomy, tubal ligation), which have been reversed. The prior procedure may affect study outcomes, and patients with both a reversed sterilization procedure and PCOS are rare enough that exclusion should not adversely affect recruitment.
   12. Subjects who have undergone a bariatric surgery procedure in the recent past (< 12 months) and are in a period of acute weight loss or have been advised against pregnancy by their bariatric surgeon.
   13. Patients with untreated poorly controlled hypertension defined as a systolic blood pressure 160 mmHg or a diastolic 100 mm Hg obtained on two measures obtained at least 60 minutes apart.
   14. Patients with known congenital adrenal hyperplasia.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — PCOS is a complex reproductive-metabolic disorder, affects 5-10% of reproductive age women and is the most common cause of anovulatory infertility.
Enrollment: 1100 (Estimated)
Dates: Start 2018-08-13 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Live birth rate | Up to 14 months
  Live birth rate defined as a delivery after ≥20 weeks gestation.

SECONDARY OUTCOMES:
Ovulation rate | Up to 4 months
  Ovulation defined as a serum progesterone level >3 ng/mL on day 21 or day 28 of the cycle.
Conception rate | Up to 4 months
  Conception defined as positive serum hCG.
Pregnancy rate | Up to 6.5 months
  Around 8-10 weeks gestation.
Pregnancy loss rate | Up to 9 months
  Pregnancy loss defined as pregnancy loss occurring from conception to 27 completed weeks of gestational age.
Follicle stimulating hormone (FSH) | Up to 4 months
  Hormonal profile
Luteinizing hormone(LH) | Up to 4 months
  Hormonal profile
Testosterone(T) | Up to 4 months
  Hormonal profile
Sex hormone-binding globulin (SHBG) | Up to 4 months
  Hormonal profile
Serum glucose concentration | Up to 4 months
  Metabolic profile
Insulin concentration | Up to 4 months
  Metabolic profile
Cholesterol | Up to 4 months
  Metabolic profile
Triglycerides (TG) | Up to 4 months
  Metabolic profile
High density lipoprotein cholesterol (HDL-C) | Up to 4 months
  Metabolic profile
Low density lipoprotein cholesterol (LDL-C) | Up to 4 months
  Metabolic profile
The scores of short form 36 (SF 36) | Up to 4 months
  SF-36 is one of questionnaires for assessments of health-related quality of life. It includes 36 items, the scores for each domain range from 0 to 100, with high scores indicating a better status.
The scores of polycystic ovary syndrome questionnaire (PCOSQ) | Up to 4 months
  PCOSQ is one of questionnaires for assessments of health-related quality of life. It concludes 26 items. Each question is associated with a 7-point scale in which 7 represents optimal function and 1 represents the poorest function.
The scores of Chinese quality of life (ChQOL) questionnaire | Up to 4 months
  ChQOL is one of questionnaires for assessments of health-related quality of life. The ChQOL is unique in that it is a health-related quality of life （HRQOL） measure specific to Traditional Chinese Medicine (TCM). ChQOL consists of 50 items ,each item is rated on a five-point Likert scale with higher scores indicating better HRQOL.
The scores of Zung Self-Rating Anxiety Scale (SAS) | Up to 4 months
  Zung SAS is one of questionnaires for symptoms of anxiety and depression. For the SAS, index score of 50 is a cut-off point for clinically significant anxiety, with higher score suggesting more serious depression.
The scores of Zung Self-reported Depression Scale (SDS) | Up to 4 months
  Zung SDS is one of questionnaires for symptoms of anxiety and depression. Index scores of 25 to 49 indicate nil depression, 50-59 indicate mild to moderate depression, 60-69 indicate moderate to severe depression, and scores over 70 indicate severe depression.
Side effect profile | Up to 14 months
  Adverse events will be categorized and percentage of patients experiencing. adverse events and serious adverse events during the treatment period will be documented.

CONTACTS AND LOCATIONS:
Overall Officials: Hongxia HX Ma, Dorctor, Study Chair — The First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- The first affiliated hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Homburg R. Management of infertility and prevention of ovarian hyperstimulation in women with polycystic ovary syndrome. Best Pract Res Clin Obstet Gynaecol. 2004 Oct;18(5):773-88. doi: 10.1016/j.bpobgyn.2004.05.006. PMID 15380146
- [Background] Thessaloniki ESHRE/ASRM-Sponsored PCOS Consensus Workshop Group. Consensus on infertility treatment related to polycystic ovary syndrome. Hum Reprod. 2008 Mar;23(3):462-77. doi: 10.1093/humrep/dem426. PMID 18308833
- [Background] Legro RS, Barnhart HX, Schlaff WD, Carr BR, Diamond MP, Carson SA, Steinkampf MP, Coutifaris C, McGovern PG, Cataldo NA, Gosman GG, Nestler JE, Giudice LC, Leppert PC, Myers ER; Cooperative Multicenter Reproductive Medicine Network. Clomiphene, metformin, or both for infertility in the polycystic ovary syndrome. N Engl J Med. 2007 Feb 8;356(6):551-66. doi: 10.1056/NEJMoa063971. PMID 17287476
- [Background] Holzer H, Casper R, Tulandi T. A new era in ovulation induction. Fertil Steril. 2006 Feb;85(2):277-84. doi: 10.1016/j.fertnstert.2005.05.078. PMID 16595197
- [Background] Franik S, Kremer JA, Nelen WL, Farquhar C, Marjoribanks J. Aromatase inhibitors for subfertile women with polycystic ovary syndrome: summary of a Cochrane review. Fertil Steril. 2015 Feb;103(2):353-5. doi: 10.1016/j.fertnstert.2014.10.016. Epub 2014 Nov 5. PMID 25455536
- [Background] Balen AH, Morley LC, Misso M, Franks S, Legro RS, Wijeyaratne CN, Stener-Victorin E, Fauser BC, Norman RJ, Teede H. The management of anovulatory infertility in women with polycystic ovary syndrome: an analysis of the evidence to support the development of global WHO guidance. Hum Reprod Update. 2016 Nov;22(6):687-708. doi: 10.1093/humupd/dmw025. Epub 2016 Aug 10. PMID 27511809
- [Background] Jedel E, Labrie F, Oden A, Holm G, Nilsson L, Janson PO, Lind AK, Ohlsson C, Stener-Victorin E. Impact of electro-acupuncture and physical exercise on hyperandrogenism and oligo/amenorrhea in women with polycystic ovary syndrome: a randomized controlled trial. Am J Physiol Endocrinol Metab. 2011 Jan;300(1):E37-45. doi: 10.1152/ajpendo.00495.2010. Epub 2010 Oct 13. PMID 20943753
- [Background] Johansson J, Redman L, Veldhuis PP, Sazonova A, Labrie F, Holm G, Johannsson G, Stener-Victorin E. Acupuncture for ovulation induction in polycystic ovary syndrome: a randomized controlled trial. Am J Physiol Endocrinol Metab. 2013 May 1;304(9):E934-43. doi: 10.1152/ajpendo.00039.2013. Epub 2013 Mar 12. PMID 23482444
- [Background] Benrick A, Kokosar M, Hu M, Larsson M, Maliqueo M, Marcondes RR, Soligo M, Protto V, Jerlhag E, Sazonova A, Behre CJ, Hojlund K, Thoren P, Stener-Victorin E. Autonomic nervous system activation mediates the increase in whole-body glucose uptake in response to electroacupuncture. FASEB J. 2017 Aug;31(8):3288-3297. doi: 10.1096/fj.201601381R. Epub 2017 Apr 12. PMID 28404742
- [Background] Wu XK, Stener-Victorin E, Kuang HY, Ma HL, Gao JS, Xie LZ, Hou LH, Hu ZX, Shao XG, Ge J, Zhang JF, Xue HY, Xu XF, Liang RN, Ma HX, Yang HW, Li WL, Huang DM, Sun Y, Hao CF, Du SM, Yang ZW, Wang X, Yan Y, Chen XH, Fu P, Ding CF, Gao YQ, Zhou ZM, Wang CC, Wu TX, Liu JP, Ng EHY, Legro RS, Zhang H; PCOSAct Study Group. Effect of Acupuncture and Clomiphene in Chinese Women With Polycystic Ovary Syndrome: A Randomized Clinical Trial. JAMA. 2017 Jun 27;317(24):2502-2514. doi: 10.1001/jama.2017.7217. PMID 28655015
- [Background] Napadow V, Kaptchuk TJ. Patient characteristics for outpatient acupuncture in Beijing, China. J Altern Complement Med. 2004 Jun;10(3):565-72. doi: 10.1089/1075553041323849. PMID 15253864
- [Background] Linde K, Streng A, Jurgens S, Hoppe A, Brinkhaus B, Witt C, Wagenpfeil S, Pfaffenrath V, Hammes MG, Weidenhammer W, Willich SN, Melchart D. Acupuncture for patients with migraine: a randomized controlled trial. JAMA. 2005 May 4;293(17):2118-25. doi: 10.1001/jama.293.17.2118. PMID 15870415
- [Background] Cherkin DC, Sherman KJ, Avins AL, Erro JH, Ichikawa L, Barlow WE, Delaney K, Hawkes R, Hamilton L, Pressman A, Khalsa PS, Deyo RA. A randomized trial comparing acupuncture, simulated acupuncture, and usual care for chronic low back pain. Arch Intern Med. 2009 May 11;169(9):858-66. doi: 10.1001/archinternmed.2009.65. PMID 19433697
- [Background] Macklin EA, Wayne PM, Kalish LA, Valaskatgis P, Thompson J, Pian-Smith MC, Zhang Q, Stevens S, Goertz C, Prineas RJ, Buczynski B, Zusman RM. Stop Hypertension with the Acupuncture Research Program (SHARP): results of a randomized, controlled clinical trial. Hypertension. 2006 Nov;48(5):838-45. doi: 10.1161/01.HYP.0000241090.28070.4c. Epub 2006 Oct 2. PMID 17015784
- [Background] Moher D, Hopewell S, Schulz KF, Montori V, Gotzsche PC, Devereaux PJ, Elbourne D, Egger M, Altman DG. CONSORT 2010 explanation and elaboration: updated guidelines for reporting parallel group randomised trials. BMJ. 2010 Mar 23;340:c869. doi: 10.1136/bmj.c869. No abstract available. PMID 20332511
- [Background] MacPherson H, Altman DG, Hammerschlag R, Youping L, Taixiang W, White A, Moher D; STRICTA Revision Group. Revised STandards for Reporting Interventions in Clinical Trials of Acupuncture (STRICTA): Extending the CONSORT statement. J Evid Based Med. 2010 Aug;3(3):140-55. doi: 10.1111/j.1756-5391.2010.01086.x. PMID 21349059
- [Background] Zhao X, Ni R, Li L, Mo Y, Huang J, Huang M, Azziz R, Yang D. Defining hirsutism in Chinese women: a cross-sectional study. Fertil Steril. 2011 Sep;96(3):792-6. doi: 10.1016/j.fertnstert.2011.06.040. Epub 2011 Jul 18. PMID 21762890
- [Background] Ni RM, Mo Y, Chen X, Zhong J, Liu W, Yang D. Low prevalence of the metabolic syndrome but high occurrence of various metabolic disorders in Chinese women with polycystic ovary syndrome. Eur J Endocrinol. 2009 Sep;161(3):411-8. doi: 10.1530/EJE-09-0298. Epub 2009 Jun 19. PMID 19542239
- [Background] Balen AH, Laven JS, Tan SL, Dewailly D. Ultrasound assessment of the polycystic ovary: international consensus definitions. Hum Reprod Update. 2003 Nov-Dec;9(6):505-14. doi: 10.1093/humupd/dmg044. PMID 14714587
- [Background] Jin C, Pang R, Xu L, Wu Z, Zhao J. [Clinical rules for acupoint selection and prescription composition in treatment of polycystic ovary syndrome with acupuncture]. Zhongguo Zhen Jiu. 2015 Jun;35(6):625-30. Chinese. PMID 26480575
- [Background] Kuang H, Li Y, Wu X, Hou L, Wu T, Liu J, Ng EH, Stener-Victorin E, Legro RS, Zhang H. Acupuncture and clomiphene citrate for live birth in polycystic ovary syndrome: study design of a randomized controlled trial. Evid Based Complement Alternat Med. 2013;2013:527303. doi: 10.1155/2013/527303. Epub 2013 Aug 20. PMID 24023577
- [Derived] Franik S, Le QK, Kremer JA, Kiesel L, Farquhar C. Aromatase inhibitors (letrozole) for ovulation induction in infertile women with polycystic ovary syndrome. Cochrane Database Syst Rev. 2022 Sep 27;9(9):CD010287. doi: 10.1002/14651858.CD010287.pub4. PMID 36165742
- [Derived] Huang S, Hu M, Ng EHY, Stener-Victorin E, Zheng Y, Wen Q, Wang C, Lai M, Li J, Gao X, Wang X, Hu Z, Xia T, Hu R, Liu J, Wen X, Li S, Quan K, Liang X, Shang H, Ma H, Qiao J. A multicenter randomized trial of personalized acupuncture, fixed acupuncture, letrozole, and placebo letrozole on live birth in infertile women with polycystic ovary syndrome. Trials. 2020 Mar 4;21(1):239. doi: 10.1186/s13063-020-4154-1. PMID 32131886